CLINICAL TRIAL: NCT03813004
Title: Kinematics and Kinetics of Gait Perturbations in Young Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Łysoń (Other)
Responsible Party: Sponsor-Investigator, Barbara Łysoń, Principal Investigator, Józef Piłsudski University of Physical Education
Organization: Józef Piłsudski University of Physical Education (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DS-311
Record Dates: First submitted 2019-01-07; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Balance Disorders
Keywords: motek grail; balance; gait perturbation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young healthy adults (Experimental)
  Interventions: Diagnostic Test: Reaction for gait perturbation

INTERVENTIONS:
Diagnostic Test: Reaction for gait perturbation — Participants were subjected to four different perturbation types while walking on the treadmill:
  1. left treadmill belt deceleration for right leg toe off
  2. right treadmill belt deceleration for left leg toe off
  3. left treadmill belt acceleration for right leg heel strike
  4. right treadmill belt acceleration for left leg heel strike
  Motion analysis was conducted to analyze effect of the intervention on gait.

SUMMARY:
Investigators would like to examine, what are strategies for balance recovery in gait perturbations. Different perturbation types where used in the current study. The study involves the analysis of kinematic and kinetic parameters. Researchers hypothesize that research including young healthy adults would help to elaborate fall prevention program for seniors.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35
* female or male
* good health condition

Exclusion Criteria:

* lower limb injuries (last 6 months)
* head injuries (last 6 months)
* diseases of the vestibular system
* serious eye defects
* extreme sports athletes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Motek Grail output (joint angles) | 40 minutes
  Joint angles calculated using HBM Gait model [degrees]
Motek Grail output (joint moments) | 40 minutes
  Joint moments calculated using HBM Gait model [Newton*meter/kilogram]
Motek Grail output (ground reaction forces) | 40 minutes
  Ground reaction forces calculated using treadmill with built-in dual 6 DoF force plates and independent belts for each foot [Newtons]
Motek Grail output (centre of pressure) | 40 minutes
  Center of pressure calculated using treadmill with built-in dual 6 DoF force plates and independent belts for each foot [meters]
Body composition | 10 minutes
  Body composition using Tanita Body Composition Monitor (fat tissue percentage, muscle mass percentage, water percentage)
Range of movement | 20 minutes
  Range of movement in hip, knee and ankle joint, measured using SFTR system [degrees]
Height | 2 minutes
  Height measured in meters
Weight | 2 minutes
  Weight measured in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Józef Piłsudski University of Physical Education in Warsaw, Warsaw, Mazowsze, Poland